CLINICAL TRIAL: NCT03835039
Title: The Ability of Near Infrared Spectroscopy Monitoring During Hypothermia Treatment to Predict Brain Injury in Infants With Hypoxic Ischemic Encephalopathy
Brief Title: The Ability of NIRS to Predict Brain Injury in Hypoxic Ischemic Encephalopathy
Status: Terminated | Type: Observational
Why Stopped: Interim analysis not showing significant results
Sponsor: Albany Medical College (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 5120
Record Dates: First submitted 2019-01-18; First posted 2019-02-08 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: HIE - Perinatal Hypoxic - Ischemic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- HIE: Infants with a diagnosis of HIE
  Interventions: Device: NIRS

INTERVENTIONS:
Device: NIRS — Monitoring cerebral and perirenal perfusion using NIRS

SUMMARY:
A longitudinal study evaluating the predictive ability of near infrared spectroscopy to predict brain injury in infants with hypoxic ischemic encephalopathy. Data will be analyzed at two different time periods, at discharge and again at 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants with diagnosis at birth of HIE

Exclusion Criteria:

* none

Ages: 1 Minute to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants with diagnosis of HIE
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
MRI findings of encephalopathy | 6 days
  MRI studies will be reviewed and assessed for markers of HIE including damage to deep grey matter structures.
Neurodevelopment at 2 years of age | 2 years
  Bayleys developmental test will be used to categorize the infants' neurodevelopment at 2 years of age.

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center Neonatal Intesive Care Unit, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No